CLINICAL TRIAL: NCT06743919
Title: Adding Magnesium Sulfate or Dexmedetomidine to Bupivacaine in Oblique Subcostal Tap Block for Laparoscopic Cholecystectomy: a Randomized Double -Blind Controlled Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Zaki Mousa Sayed Mansour, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSCTAP Cholecystectomy
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Oblique Subcostal Tap Block
MeSH Terms: interventions — Magnesium Sulfate; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- group 1 (Experimental): patient will receive 20 ml bupivacaine 0.25% plus 500 mg magnesium sulfate in 5ml normal saline on both sides.
  Interventions: Drug: Magnesium sulfate 50% - 1g/h; Drug: Bupivacaine
- group 2 (Experimental): patients will receive 20 ml bupivacaine 0.25% plus o .5 microg per kg dexmedetomidine in 5 ml normal saline on both sides.
  Interventions: Drug: dexmedetomidine 0.5 µg/kg IV; Drug: Bupivacaine
- group 3 (Placebo Comparator): patients will receive 20 ml bupivacaine 0.25% plus 5 ml normal saline on both sides.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Magnesium sulfate 50% - 1g/h — magnesium sulfate group 20 ml bupivacaine 0.25% plus 500 mg magnesium sulfate in 5ml normal saline on both sides.
  Arms: group 1
Drug: dexmedetomidine 0.5 µg/kg IV — dexmedetomidine group 20 ml bupivacaine 0.25% plus o .5 microg per kg dexmedetomidine in 5 ml normal saline on both sides.
  Arms: group 2
Drug: Bupivacaine — 20 ml bupivacaine 0.25% plus 5 ml normal saline on both sides.

SUMMARY:
Laparoscopic cholecystectomy (LC) is one of the commonly performed surgical procedures associated with a moderate degree of postoperative pain especially on the 1st postoperative day. Adequate postoperative analgesia allows early patient ambulation, decreases analgesic requirements, and hospital stay. Moreover, it has been hypothesized that intense acute pain after LC may predict development of chronic pain (e.g., post laparoscopic cholecystectomy syndrome). So, aggressive perioperative analgesia is needed.

the aim of the study is To compare the analgesic effect of magnesium sulfate combined with bupivacaine versus bupivacaine combined dexmedetomidine via OSCTAB block on postoperative pain control for 24 hours in patients scheduled for LC.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block is a recent analgesic technique with efficacy in perioperative pain therapy for LC. It involves the infusion of local anesthetic into the fascial plane of the abdominal wall.

Oblique subcostal transversus abdominis plane (OSCTAP) block is an US-guided regional anesthesia technique that anesthetizes the nerves of the lower and upper anterior abdominal wall, specifically from T6 to L1. There weren't enough studies in the literature evaluating the OSCTAP block for pain management after LC.

Rafi et al and McDonnell et al were first to describe this novel abdominal field block. They described an anatomical landmark technique and provided evidence of blockade to the mid/lower thoracic and upper lumbar spinal nerves as they travelled in the fascial plane between the transversus abdominis (TA) and internal oblique (IO) muscles.

The OSCTAB block provides more effective analgesia than other TAP blocks. Numerous regional anesthetic adjuvants.

such as dexmedetomidine, clonidine, epinephrine, dexamethasone, and magnesium sulphate (MgSO4) are usually combined with enhancement of analgesic efficacy.

Recently, these adjuvants added to LA solution for prolonging the effect of TAP block with promising results.

ELIGIBILITY:
Inclusion Criteria:

* • Patients programmed for elective LC.

  * American society of anesthesiologists (ASA) physical state I or II.
  * Age over 18 years and less than 60 years old.
  * Patients of both sex are included in the study.

Exclusion Criteria:

* •Patient refusal

  * Known hypersensitivity to the study drugs.
  * Body Mass Index > 40 kg/m2.
  * Inability to accurately describe postoperative pain to investigators.
  * Opioid tolerance or dependence.
  * Preexisting history of chronic pain.
  * History of renal, liver, cardiac, neuropsychiatric disorder problems.
  * Bleeding or coagulation abnormality.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
post operative ( NRS score | 24 hours
  analgesic effect of OSCTAB block on postoperative pain control according to (NRS) for 24 hours in patients scheduled for LC.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun C, He Z, Feng B, Huang Y, Liu D, Sun Z. Effect of Intraperitoneal Instillation of Dexmedetomidine With Local Anesthetics in Laparoscopic Cholecystectomy: A Systematic Review and Meta-analysis of Randomized Trials. Surg Laparosc Endosc Percutan Tech. 2024 Apr 1;34(2):222-232. doi: 10.1097/SLE.0000000000001262. PMID 38359350
- [Background] Lee TH, Barrington MJ, Tran TM, Wong D, Hebbard PD. Comparison of extent of sensory block following posterior and subcostal approaches to ultrasound-guided transversus abdominis plane block. Anaesth Intensive Care. 2010 May;38(3):452-60. doi: 10.1177/0310057X1003800307. PMID 20514952
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Background] Hutchins J, Delaney D, Vogel RI, Ghebre RG, Downs LS Jr, Carson L, Mullany S, Teoh D, Geller MA. Ultrasound guided subcostal transversus abdominis plane (TAP) infiltration with liposomal bupivacaine for patients undergoing robotic assisted hysterectomy: A prospective randomized controlled study. Gynecol Oncol. 2015 Sep;138(3):609-13. doi: 10.1016/j.ygyno.2015.06.008. Epub 2015 Jun 6. PMID 26056753
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Bisgaard T, Rosenberg J, Kehlet H. From acute to chronic pain after laparoscopic cholecystectomy: a prospective follow-up analysis. Scand J Gastroenterol. 2005 Nov;40(11):1358-64. doi: 10.1080/00365520510023675. PMID 16334446
- [Background] Petersen PL, Stjernholm P, Kristiansen VB, Torup H, Hansen EG, Mitchell AU, Moeller A, Rosenberg J, Dahl JB, Mathiesen O. The beneficial effect of transversus abdominis plane block after laparoscopic cholecystectomy in day-case surgery: a randomized clinical trial. Anesth Analg. 2012 Sep;115(3):527-33. doi: 10.1213/ANE.0b013e318261f16e. Epub 2012 Jul 4. PMID 22763903